CLINICAL TRIAL: NCT00706056
Title: A New View of Normal Tension Glaucoma: Autoregulation and Systemic Blood Pressure
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Mary E. Charlson, MD, Principal Investigator, Weill Medical College of Cornell University
Other Study IDs: 0712009565
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Normal Tension Glaucoma
MeSH Terms: conditions — Low Tension Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to determine whether systemic blood pressure in the body is related to the development and progression of normal tension glaucoma in the eye. The study aims to clarify whether subjects with episodes of hypotension (low blood pressure) at night are at increased risk for sight loss and the development of normal tension glaucoma.

DETAILED DESCRIPTION:
Glaucoma is an eye disease that leads to damage of the optic nerve, visual field loss and can progress to blindness. Traditionally, glaucoma and its treatment have been closely linked to intraocular pressures. In normal tension glaucoma, damage to the optic nerve occurs without any increase in intraocular pressure. Normal tension glaucoma most often occurs in the elderly and can lead to loss of sight and significant disability. Subjects with progressive visual field loss are often a highly motivated group of subjects, ready to take an active part in the treatment of their condition. Investigating the risk factors that contribute to the development of normal-tension glaucoma may shed light on the progression of the disease.

Subjects with normal tension glaucoma will have their demographic and clinical characteristics recorded and their eyes examined at baseline, 6-months and 12 months. Subjects will wear an external blood pressure cuff for 48 hours that will record blood pressure every 30 minutes. This same blood pressure recording procedure will be performed at baseline, at 6 months, and at 12 months. At these same time intervals, visual fields will also be measured, as per routine clinical care, by the treating ophthalmologist. The results of the visual field testing will be recorded. The primary outcome of the study will be visual field abnormalities and their relationship to dips in systemic blood pressure. Results will be published and will be used as a base for future projects that may impact treatment and the understanding of risk factors of normal tension glaucoma.

ELIGIBILITY:
Inclusion Criteria:

1. The IOP must be less than or equal to 21 mmHg without treatment and must have never been higher than 24 mmHg, without treatment.
2. Gonioscopically open angles.
3. Typical glaucomatous optic disc changes, including: rim thinning, cupping, rim notching, disc hemorrhage, nerve fiber layer defect, vertical cup/disc asymmetry ≥0.2.
4. A reproducible visual field defect must have been demonstrated on at least three prior visual fields, as observed using standard automated perimetry with Swedish Interactive Threshold Algorithm (SITA-STANDARD) from the Humphrey Visual Field Analyzer using the 24-2 test pattern.
5. There must have been progression of glaucomatous loss with the past 36 months, specifically, two or more adjacent non-peripheral points changed by 10dB relative to the average baseline value for the points, confirmed by two subsequent fields.

Exclusion Criteria:

1. Subjects with a visual field defect attributable to conditions other than glaucoma, such as a history of intra-cranial or ENT mass lesion.
2. Occludable narrow angles.
3. Subjects with intermittent elevation of intraocular pressure associated with another form of glaucoma, including intermittent angle closure, inflammatory glaucoma, old pigmentary glaucoma, psedoexfoliation or uveitis.
4. Subjects who cannot complete follow-up testing every six months for any reason.
5. Subjects who are unable to provide informed consent or who refuse or whose physicians do not wish for the subjects to participate for any reason.

Ages: 21 Years to 101 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Normal Tension Glaucoma
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome of the study will be visual field abnormalities and their relationship to dips in systemic blood pressure. | baseline, 6-months and 12-months

CONTACTS AND LOCATIONS:
Overall Officials: Mary E. Charlson, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - Glaucoma Associates of New York/New York Eye and Ear Infirmary, New York, New York
  - The New York Presbyterian Hospital-Weill Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No
No Plan to Share IPD